CLINICAL TRIAL: NCT01372995
Title: High-Dose Vitamin D and Antimicrobial Peptide Expression in Lung Failure
Brief Title: Vitamin D in Ventilated ICU Patients
Acronym: R21 HL-110044
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Greg S. Martin, M.D., M.Sc., Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00049610
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Respiratory Failure
Keywords: critical care; nosocomial infection; antiAntimicrobial peptide expression; LL-37; hBD-2; cathelicidin; microbial peptide
MeSH Terms: conditions — Respiratory Insufficiency; Cross Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Enteral vitamin D3 50,000 IU (Experimental): An arm where subjects receive 50,000 IU of Vitamin D for 5 days.
  Interventions: Drug: Enteral Vitamin D3 50,000 IU
- Enteral Vitamin D3 100,000 IU (Experimental): Arm where subjects receive 100,000 IU of Vitamin D for 5 days
  Interventions: Drug: Enteral Vitamin D3 100,000IU
- Inactive Substance (Placebo Comparator): Arm where patients receive inactive substance for 5 days.
  Interventions: Other: Inactive substance

INTERVENTIONS:
Drug: Enteral Vitamin D3 50,000 IU — Enteral Vitamin D3 50,000IU x 5 days (total dose 250,000IU)
  Arms: Enteral vitamin D3 50,000 IU
Drug: Enteral Vitamin D3 100,000IU — Enteral Vitamin D3 100,000IU over 5 days (total 500,000IU)
  Arms: Enteral Vitamin D3 100,000 IU
Other: Inactive substance — Inactive substance given enterally for 5 days.
  Arms: Inactive Substance

SUMMARY:
The increasing rate of hospital-acquired infection and antibiotic resistance are major causes of prolonged ICU stay and death in hospitalized patients. The enormous impact of ICU-related infection demands the need for cost-effective therapies that can be rapidly implemented to improve patient immune response to control infection. Unfortunately, little high-quality comparative effectiveness research has been performed on micronutrient treatment regimens as methods to decrease hospital-acquired infection in critically ill patients. Critically ill medical and surgical patients have an extremely high prevalence of vitamin D insufficiency.

We will perform a rigorous, double-blind, randomized, controlled, pilot clinical trial in ventilator-dependent ICU patients to test the clinical/metabolic safety and efficacy of two doses of oral high-dose vitamin D3 therapy versus standard therapy (no supplemental vitamin D). The primary endpoint is to test whether high-dose regimens [either 50,000 or 100,000 international units (IU) of enteral vitamin D3 given daily for 5 consecutive days (total dose = 250,000 or 500,000 IU, respectively) increase plasma 25(OH)D concentrations into a desirable range (> 30 ng/mL).

DETAILED DESCRIPTION:
1. We will evaluate, over 12 weeks, the safety and efficacy of two high-dose vitamin D3 regimens in severely ill ICU patients. Vitamin D or placebo ( depending on study arm) will be given sequentially in divided doses for 5 days
2. We will explore whether these vitamin D regimens are capable of increasing the production of key antimicrobial peptides LL-37 and hBD-2 ( substances produced by our bodies to fight infections), in both the blood and in lung.
3. We will determine whether a higher vitamin D level in the blood is associated with a decrease in hospital infection rates and other complications in high-risk ICU patients with respiratory failure.

Study Design:

Enrollment goal is 36 patients. Once consent is obtained subjects will be randomly assigned to one of three study groups. Each group consists of 12 patients with enteral access ; a placebo arm, an arm where subjects receive 50,000 IU of Vitamin D for 5 days, and a third arm where subjects receive 100,000 IU of Vitamin D for 5 days.

Methods: Baseline blood samples (25-hydroxyvitamin D, vitamin D binding protein, ionized calcium, LL-37,and hBD-2) will be taken on study day 7,14,21,28,84 days. On study day 1 and 8, LL-37, hBD-2, cathelicidin from BAL fluid will also be analyzed. Patients will be given either placebo, Vitamin D3 50,000 IU x 5 days (total 250,000 IU) or Vitamin D3 100,000 IU x 5 days (total 500,000 IU) with an intention to treat model. Baseline data on the patients including demographic, laboratory, documented infections, severity illness score (APACHE II) and organ dysfunction score (SOFA) will be collected. ELISA assay on the serum and BAL will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care in an intensive care unit (ICU)
* Age greater than 18 years
* Expected to require mechanical ventilation for at least 72 hours after entry
* Expected to survive and remain in the ICU for at least 96 hours after study entry
* To enable delivery of study drug, the subject has enteral access in place and is deemed able to tolerate enteral drug administration

Exclusion Criteria:

* Inability to obtain or declined informed consent from the subject and/or legally authorized representative
* Pregnancy
* Ongoing shock
* Current hypercalcemia (albumin-corrected serum calcium > 10.8 mg/dL or ionized calcium > 5.2 mg/dL)
* History of therapy with high-dose vitamin D to treat vitamin D deficiency within previous 6 months
* History of disorders associated with hypercalcemia; history of cancer with history of hypercalcemia within the past 1 year, hyperparathyroidism, sarcoidosis, nephrolithiasis]
* Chronic renal dysfunction requiring chronic dialysis
* Known history of cirrhosis
* History of AIDS
* The patient has received any investigational drug within 60 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Martin, MD, MSc, Principal Investigator — Emory University; Thomas Ziegler, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

REFERENCES:
- [Background] Tejada Artigas A, Bello Dronda S, Chacon Valles E, Munoz Marco J, Villuendas Uson MC, Figueras P, Suarez FJ, Hernandez A. Risk factors for nosocomial pneumonia in critically ill trauma patients. Crit Care Med. 2001 Feb;29(2):304-9. doi: 10.1097/00003246-200102000-00015. PMID 11246310
- [Background] Winther B, Greve JM, Gwaltney JM Jr, Innes DJ, Eastham JR, McClelland A, Hendley JO. Surface expression of intercellular adhesion molecule 1 on epithelial cells in the human adenoid. J Infect Dis. 1997 Aug;176(2):523-5. doi: 10.1086/517280. PMID 9237723
- [Background] Urashima M, Segawa T, Okazaki M, Kurihara M, Wada Y, Ida H. Randomized trial of vitamin D supplementation to prevent seasonal influenza A in schoolchildren. Am J Clin Nutr. 2010 May;91(5):1255-60. doi: 10.3945/ajcn.2009.29094. Epub 2010 Mar 10. PMID 20219962
- [Background] Manaseki-Holland S, Qader G, Isaq Masher M, Bruce J, Zulf Mughal M, Chandramohan D, Walraven G. Effects of vitamin D supplementation to children diagnosed with pneumonia in Kabul: a randomised controlled trial. Trop Med Int Health. 2010 Oct;15(10):1148-55. doi: 10.1111/j.1365-3156.2010.02578.x. Epub 2010 Aug 17. PMID 20723187
- [Background] Yim S, Dhawan P, Ragunath C, Christakos S, Diamond G. Induction of cathelicidin in normal and CF bronchial epithelial cells by 1,25-dihydroxyvitamin D(3). J Cyst Fibros. 2007 Nov 30;6(6):403-10. doi: 10.1016/j.jcf.2007.03.003. Epub 2007 Apr 27. PMID 17467345
- [Background] De Smet K, Contreras R. Human antimicrobial peptides: defensins, cathelicidins and histatins. Biotechnol Lett. 2005 Sep;27(18):1337-47. doi: 10.1007/s10529-005-0936-5. PMID 16215847
- [Background] Barlow PG, Beaumont PE, Cosseau C, Mackellar A, Wilkinson TS, Hancock RE, Haslett C, Govan JR, Simpson AJ, Davidson DJ. The human cathelicidin LL-37 preferentially promotes apoptosis of infected airway epithelium. Am J Respir Cell Mol Biol. 2010 Dec;43(6):692-702. doi: 10.1165/rcmb.2009-0250OC. Epub 2010 Jan 22. PMID 20097832
- [Background] Jeng L, Yamshchikov AV, Judd SE, Blumberg HM, Martin GS, Ziegler TR, Tangpricha V. Alterations in vitamin D status and anti-microbial peptide levels in patients in the intensive care unit with sepsis. J Transl Med. 2009 Apr 23;7:28. doi: 10.1186/1479-5876-7-28. PMID 19389235
- [Derived] Han JE, Jones JL, Tangpricha V, Brown MA, Brown LAS, Hao L, Hebbar G, Lee MJ, Liu S, Ziegler TR, Martin GS. High Dose Vitamin D Administration in Ventilated Intensive Care Unit Patients: A Pilot Double Blind Randomized Controlled Trial. J Clin Transl Endocrinol. 2016 Jun;4:59-65. doi: 10.1016/j.jcte.2016.04.004. Epub 2016 May 5. PMID 27419080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from critical care units at three hospitals in Atlanta, Georgia. 658 patients were assessed for eligibility, of these 562 did not meet inclusion and exclusion criteria. 65 eligible patients declined to participate while 31 gave informed consent and were randomized to one of the three study arms.
Groups:
- Placebo: Participants randomized to receive an inactive substance administered enterally for 5 days
- 250,000 IU of Vitamin D3: Participants randomized to receive 50,000 IU of Vitamin D3 per day for 5 days, for a total dose of 250,000 IU administered enterally
- 500,000 IU of Vitamin D3: Participants randomized to receive 100,000 IU per day of Vitamin D3 for 5 days, for a total dose of 500,000 administered enterally
Period: Overall Study
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Started | 10 | 10 | 11 (One participant was transferred to comfort care prior to completing the intervention.)
Completed | 10 | 9 | 10 (The transferred participant was included in the intent to treat analyses.)
Not Completed | 0 | 1 | 1
Not completed — Spouse withdrew participant from study | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The participant randomized to the 250,000 IU of Vitamin D3 study arm, whose spouse withdrew consent to participate in the study, is not represented in the Baseline Analysis Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3 | Total
Number analyzed (Participants) | 10 | 9 | 11 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 4 | 14
  >=65 years | 5 | 4 | 7 | 16
Gender [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 11
  Male | 6 | 5 | 8 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 4 | 7 | 3 | 14
  Caucasian | 5 | 2 | 8 | 15
  American Indian/Alaskan | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 11 | 30
Vitamin D at baseline [Number; unit: participants]
  Deficient (<20 ng/mL) | 5 | 3 | 5 | 13
  Insufficient (20-30 ng/mL) | 3 | 4 | 5 | 12
  Sufficient (>30 ng/mL) | 2 | 2 | 1 | 5
Coronary Artery Disease [Number; unit: participants]
  Coronary Artery Disease Present | 1 | 2 | 7 | 10
  No Coronary Artery Disease | 9 | 7 | 4 | 20
Congestive Heart Failure [Number; unit: participants]
  Congestive Heart Failure Present | 1 | 2 | 5 | 8
  No Congestive Heart Failure | 9 | 7 | 6 | 22
Diabetes [Number; unit: participants]
  Diabetes Present | 4 | 1 | 2 | 7
  No Diabetes | 6 | 8 | 9 | 23
Chronic Obstructive Pulmonary Disease (COPD) [Number; unit: participants]
  COPD Present | 2 | 1 | 4 | 7
  No COPD | 8 | 8 | 7 | 23
Asthma [Number; unit: participants]
  Asthma Present | 1 | 1 | 0 | 2
  No Asthma | 9 | 8 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Plasma 25(OH)D Concentration >30ng/mL at Baseline
Description: The number of participants with a plasma 25(OH)D concentration in the desirable range (defined as greater than 30 ng/mL) at the baseline measurement.
Time Frame: Baseline
Population: Blood samples were obtained every 7 days while participants remained hospitalized. Follow up discontinued once the participant was discharged from the hospital. At the baseline time point, 10 patients were randomized to the placebo arm, 9 to the arm receiving 250,000 IU of Vitamin D3, and 11 to the arm receiving 500,000 of Vitamin D3.
Measure: Number; unit: participants
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 10 | 9 | 11
participants | 2 | 2 | 1

2. Primary Outcome: Number of Participants With Plasma 25(OH)D Concentration >30ng/mL at Day 7
Description: The number of participants with a plasma 25(OH)D concentration in the desirable range (defined as greater than 30 ng/mL) at the Day 7 measurement.
Time Frame: Day 7
Population: Blood samples were obtained every 7 days while participants remained hospitalized. Follow up discontinued once the participant was discharged from the hospital. The number of participants analyzed at each time point decreased over the course of the study as participants were discharged from the hospital.
Measure: Number; unit: participants
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 9 | 6 | 9
participants | 2 | 4 | 9

3. Primary Outcome: Number of Participants With Plasma 25(OH)D Concentration >30ng/mL at Day 14
Description: The number of participants with a plasma 25(OH)D concentration in the desirable range (defined as greater than 30 ng/mL) at the Day 14 measurement.
Time Frame: Day 14
Population: Blood samples were obtained every 7 days while participants remained hospitalized. Follow up discontinued once the participant was discharged from the hospital. The number of participants analyzed for each time point decreased over the course of the study as participants were discharged from the hospital.
Measure: Number; unit: participants
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 8 | 6 | 5
participants | 2 | 5 | 5

4. Primary Outcome: Number of Participants With Plasma 25(OH)D Concentration >30ng/mL at Day 21
Description: The number of participants with a plasma 25(OH)D concentration in the desirable range (defined as greater than 30 ng/mL) at the Day 21 measurement.
Time Frame: Day 21
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 4 | 4 | 2
participants | 1 | 3 | 2

5. Primary Outcome: Number of Participants With Plasma 25(OH)D Concentration >30ng/mL at Day 28
Description: The number of participants with a plasma 25(OH)D concentration in the desirable range (defined as greater than 30 ng/mL) at the Day 28 measurement.
Time Frame: Day 28
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 3 | 2 | 1
participants | 0 | 2 | 1

6. Primary Outcome: Number of Participants With Plasma 25(OH)D Concentration >30ng/mL at Day 84
Description: The number of participants with a plasma 25(OH)D concentration in the desirable range (defined as greater than 30 ng/mL) at the Day 84 measurement.
Time Frame: Day 84
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 1 | 2 | 1
participants | 1 | 0 | 0

7. Secondary Outcome: Change in Plasma LL-37 Levels
Description: Plasma LL-37 was measured at Baseline, Day 7 and Day 14.
Time Frame: Baseline, Day 7, Day 14
Population: For the Day 14 analysis there were 8 participants in the Placebo arm, 6 participants in the 250,000 of Vitamin D arm, and 5 participants in the 500,000 of Vitamin D arm.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 8 | 6 | 5
ng/mL
  Day 7 Compared to Baseline | -3.8 [-18.9 to 26.9] | 6.0 [-13.4 to 39.2] | -13.5 [-48.4 to 37.4]
  Day 14 Compared to Baseline | 1.1 [-24.6 to 10.8] | -12.3 [-36.1 to 8.1] | -6.0 [-27.3 to 2.0]

8. Secondary Outcome: Duration of Time on Ventilator
Description: The number of days spent on mechanical ventilation was collected for all study participants and the average number of days for each study arm is reported.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 10 | 9 | 11
days | 20 (15) | 12 (10) | 14 (10)

9. Secondary Outcome: Duration of Time in Intensive Care Unit (ICU)
Description: The number of days spent in the intensive care unit (ICU) was collected for each participant and the average number of days for each study arm is reported.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 10 | 9 | 11
days | 23 (14) | 17 (14) | 15 (10)

10. Secondary Outcome: Duration of Time in Hospital
Description: The number of days that each participant spent in the hospital was collected and the average number of days for each study arm is reported.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 10 | 9 | 11
days | 36 (19) | 25 (14) | 18 (11)

11. Secondary Outcome: Change in Sequential Organ Failure Assessment (SOFA) Score
Description: Change in Sequential Organ Failure Assessment (SOFA) score between Baseline and Day 7. The Sequential Organ Failure Assessment (SOFA) score is a mortality prediction score that is based on the degree of dysfunction of 6 organ systems (respiratory, nervous, cardiovascular, liver, coagulation, and kidneys). A score ranges from 0-24. 0 (normal) to 4 (high degree of dysfunction) is given for each organ system, with a higher score indicating greater severity. A score of 0-6 is associated with a mortality rate of less than 10% while a score between 16 and 24 is associated with a greater than 90% mortality rate. Scores decreasing between the Baseline and Day 7 measurements are represented as negative values for the change in SOFA score.
Time Frame: Baseline, Day 7
Population: SOFA score obtained daily while in the ICU. The portion of the study participants included in the analysis of the change in SOFA score between Baseline and Day 7 is limited to participants having values for both time points..
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 10 | 7 | 9
units on a scale | -2 (3) | -3 (3) | -2 (3)

12. Secondary Outcome: Number of Hospital Acquired Infections
Description: The number of study participants who had a hospital acquired infection.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 10 | 9 | 11
participants | 3 | 3 | 2

13. Secondary Outcome: Number of Hospital Mortality Cases
Description: The number of study participants who died while in the hospital was collected.
Time Frame: 12 weeks
Population: The number of participants in the hospital mortality analysis for the arm receiving 500,000 IU of Vitamin D3 was 10, rather than 11.
Measure: Number; unit: participants
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 10 | 9 | 10
participants | 1 | 0 | 1

14. Secondary Outcome: Day 84 Mortality
Description: The number of participants who died prior to the end of the study (Day 84) was collected.
Time Frame: Day 84
Population: The number of participants in the hospital mortality analysis for the arm receiving 500,000 IU of Vitamin D3 was 10, rather than 11, as one participant withdrew.
Measure: Number; unit: participants
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Number analyzed (Participants) | 10 | 9 | 10
participants | 2 | 1 | 4

ADVERSE EVENTS:
Time Frame: Data regarding serious adverse events and non-serious adverse events were collected from the start of treatment until 30 days after study drug discontinuation (35 days in total). Ongoing events were monitored until resolution.
Description: As critically ill study patients are known to have a high morbidity and mortality rate, no adverse events specifically due to the study drug were expected. The clinical course of every participant was monitored to record any unexpected adverse events and all serious adverse events (SAEs). SAEs were defined as death, rehospitalization or reoperation within 30 days, cardiopulmonary arrest, pulmonary aspiration during feeding tube administration, new cancer diagnosis, and congenital anomalies.
Arm/Group | Placebo | 250,000 IU of Vitamin D3 | 500,000 IU of Vitamin D3
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/9 | 2/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | 250,000 IU of Vitamin D3 (N=9) | 500,000 IU of Vitamin D3 (N=11)
Re-hospitalization (General disorders) | 1 (1) | 1 (1) | 0 (0) — Re-hospitalization within 30 days of study drug discontinuation
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) — Death within 30 days of study drug discontinuation
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Cardiopulmonary arrest

LIMITATIONS AND CAVEATS:
Limitations to generalizability of this pilot study include the small sample size and imbalances in chronic conditions between treatment arms at study entry.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes